CLINICAL TRIAL: NCT02670681
Title: Effects of Different Intensities of Aerobic Exercise on Blood Pressure Levels of Resistant Hypertensive Subjects
Brief Title: Effects of Aerobic Exercise on Blood Pressure Levels of Resistant Hypertensive Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Leone Severino do Nascimento, Leone Severino do Nascimento, Universidade Federal da Paraíba, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0602/14
Record Dates: First submitted 2016-01-28; First posted 2016-02-02 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Hypertension; Resistant Hypertension
Keywords: Exercise; Aerobic Exercise
MeSH Terms: conditions — Hypertension; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aerobic Exercise Mild Intensity (Active Comparator): The subjects engage in aerobic exercise training (8 weeks) of mild intensity (continuous). The intensity is controlled by a corresponding heart rate at anaerobic threshold.
  Interventions: Behavioral: Aerobic Exercise Training
- Aerobic Exercise Moderate Intensity (Active Comparator): The subjects engage in aerobic exercise training (8 weeks) of moderate intensity (continuous). The intensity is controlled by a corresponding heart rate between anaerobic threshold and respiratory compensation point.
  Interventions: Behavioral: Aerobic Exercise Training
- Aerobic Exercise High Intensity (Active Comparator): The subjects engage in aerobic exercise (8 weeks) of high intensity interval training. The intensity is controlled by a corresponding heart rate above respiratory compensation point.
  Interventions: Behavioral: Aerobic Exercise Training

INTERVENTIONS:
Behavioral: Aerobic Exercise Training — 8 week of aerobic exercise training in different intensities.

SUMMARY:
The aim of this intervention study is to evaluate the acute and chronic effects of different intensity (mild, moderate and high intensity) of aerobic exercise on blood pressure levels of subjects classified as resistant hypertension. Resistant hypertensives subjects aged 40 to 70, men or women with body mass index lower that 40 kg/m² are recruited and subjected in acute phase in three sessions of aerobic exercise: mild, moderate, high intensity; and session control. After, the subjects will be randomly allocated into four intervention groups: mild intensity group, moderate intensity group, high intensity group and control group. In both phases, the subjects have blood pressure data recorded by ambulatory blood pressure monitoring, for clinic and ambulatory analysis. In addition, continuously be registered biological signs of blood pressure (finometer), electrocardiogram (DII derivation) and blood flow (venous occlusion plethysmography) for analysis of cardiac autonomic modulation, vascular autonomic modulation, baroreflex sensitivity, vasodilator response and peripheral vascular resistance.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 70 years
* Men or women
* Body mass index under 40 kg / m²
* Able to participate in exercise
* No regular physically active in the last 4 months

Exclusion Criteria:

- Smoking; with history of ischemic stroke or hemorrhagic; or coronary heart disease; or obstructive pulmonary disease or chronic restrictive; or diabetes mellitus; or chronic atrial fibrillation.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-10 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Systolic, diastolic and media blood pressure | Pre and post-intervention (8 weeks)
  Control in blood pressure levels, assess by the method of Ambulatory Blood Pressure Monitoring (ABPM), from decrease of blood pressure in measurements pre and post-intervention with physical exercise.

SECONDARY OUTCOMES:
Vasodilator Response | Pre and post-intervention (8 weeks)
  Improve in vasodilator response, assess by the method of venous occlusion plethysmography, verified by increased of 10% in blood flow in measurements pre and post-intervention with physical exercise.
  Improve in vasodilator response, assess by the method of venous occlusion plethysmography, verified by incresead of 10% in blood flow in measurements pre and post-intervention with physical exercise.
Autonomic Modulation | Pre and post-intervention (8 weeks)
  Improve in autonomic modulation, assess by spectral analysis, verified by increased of 10% parasympathetic modulation and/or by decrease of 10% of sympathetic modulation in measurements pre and post-intervention with physical exercise.
Baroreflex Sensitivity | Pre and post-intervention (8 weeks)
  Improve in baroreflex sensitivity, assess by alpha index, verified by increased of 10% in sensitivity in measurements pre and post-intervention with physical exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Training Study Laboratory Applied to Health; Departament of Physical Education, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No
Individual data are not the most important points of this study, but the results for the overall sample (external validity of the results found).

REFERENCES:
- [Derived] Nascimento LS, Santos AC, Lucena J, Silva L, Almeida A, Brasileiro-Santos MS. Acute and chronic effects of aerobic exercise on blood pressure in resistant hypertension: study protocol for a randomized controlled trial. Trials. 2017 Jun 2;18(1):250. doi: 10.1186/s13063-017-1985-5. PMID 28578691